CLINICAL TRIAL: NCT06415253
Title: Comparison of ARISCAT Score and Post-operative Pulmonary Complication Rate in Percutaneous Nephrolithotomy Cases: The Effect of Prone Position and Endoscopic Intervention
Brief Title: Comparison of ARISCAT Score and Post-operative Pulmonary Complication Rate in Percutaneous Nephrolithotomy
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, ahmet kaya, assistant professor, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: MAIEAH630003
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Complications; Nephrolithotomy, Percutaneous
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had undergone Percutaneous Nephrolithotomy

SUMMARY:
Postoperative pulmonary complications are relatively common in all age groups and are closely related to increased costs, morbidity and mortality in the postoperative period. In recent years, various risk indices have been developed for preoperative evaluation to predict postoperative pulmonary complications, such as the American Society of Anaesthesiologists Physical Status Classification (ASA), the Assessment of Respiratory Risk in Surgical Patients in Catalonia (ARISCAT). The ARISCAT score has demonstrated promising results in identifying patients at higher risk for pulmonary complications. The ARISCAT risk index is derived from multiple variables, including age, oxygen saturation, previous respiratory tract infections, anaemia, abdominal or thoracic surgery, operative time, and emergency surgery. The ARISCAT risk index is used to predict respiratory failure, bronchospasm, respiratory tract infections, atelectasis, pneumothorax, pleural effusion, and aspiration pneumonia.

Percutaneous nephrolithotomy (PNL) is a type of operation performed endoscopically in a prone position in cases of kidney stones that cannot be broken by extracorporeal shockwave lithotripsy (ESWL) and/or cannot be removed by ureterocystoscopy. The prone position is one of the positions that limits lung capacity and respiratory function. The objective of this study was to assess the relationship between the ARISCAT score in patients undergoing PNL and the occurrence of pulmonary complications in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-III patients
* Patients who undergone of Percutaneous Nephrolithotomy procedure

Exclusion Criteria:

* Patients with any liver and/or kidney failure
* Obese patients (body mass index (BMI) 30 and above)
* Trauma patients
* Cancer patients
* American Society of Anesthesiologists (ASA) IV patients
* Cardiac arrhythmia, implanted pacemakers
* A history of chronic pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included 50 ASA I-III patients aged between 18 and 80 years who were about to undergo percutaneous nephrolithotomy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
rate of pulmonary complication | The postoperative period in the first 24 hours
  rate of pulmonary complication such as respiratory failure, bronchospasm, atelectasis, pneumothorax, pleural effusion, or aspiration pneumonia.
rate of lung infection | The postoperative period in the first 72 hours
  rate of pneumonia (bacterial or virutic)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Turkey Sanliurfa Mehmet Akif Inan Training and Research Hospital, Sanliurfa, Turkey (Türkiye)